CLINICAL TRIAL: NCT05783037
Title: Growth, Tolerance, and Safety Study of Healthy Term Infants Consuming a New Organic Cow's Milk-Based Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bobbie Baby, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BB-01
Record Dates: First submitted 2023-03-16; First posted 2023-03-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Healthy Growth
Keywords: Organic; Bobbie; Bobbie Baby; Weight; Growth; Breastfeeding; Infant Formula; Growth and Tolerance
MeSH Terms: conditions — Body Weight; Breast Feeding

STUDY DESIGN:
Intervention Model Description: A decentralized, randomized, controlled trial of healthy term breastfed and formula-fed infants for 16 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- New Organic Infant Formula (Experimental): New organic infant formula for healthy term infants
  Interventions: Other: New Organic Infant Formula
- Commercial Organic Infant Formula (Active Comparator): Commercially available organic infant formula for healthy term infants
  Interventions: Other: Commercial Organic Infant Formula
- Breastfed Reference Group (No Intervention): Breastmilk

INTERVENTIONS:
Other: New Organic Infant Formula — New organic infant formula fed daily ad libitum
  Arms: New Organic Infant Formula
Other: Commercial Organic Infant Formula — Commercially available organic infant formula fed daily ad libitum
  Arms: Commercial Organic Infant Formula

SUMMARY:
The goal of this study is to demonstrate that healthy term babies who are fed Bobbie's study formula grow at the same rate as those fed with an existing cow's milk formula. Breastfeeding is the ultimate reference for infant nutrition. Therefore, this study also includes a group of breastfed babies for additional comparison.

DETAILED DESCRIPTION:
This is a 16 week, double-blind, randomized, controlled trial designed to demonstrate that a new infant formula for term infants supports age-appropriate growth. The study has been designed in accordance with Good Clinical Practice guidelines and the requirements of the Code of Federal Regulations 21 CFR 106.96

ELIGIBILITY:
Inclusion Criteria:

* Healthy gestational term (≥ 37 wks; ≤ 41 wks and 6 days)
* Birth weight of ≥ 2,500 g and ≤ 4,500 g
* Postnatal age ≤ 11 days at time of enrollment
* Singleton
* Caregiver who has previously decided to exclusively feed infant formula or exclusively breastfeed and is willing to continue with current feeding method throughout the study (breastfeeding or formula feeding)
* Caregiver willing to conform to protocol requirements (e.g. measuring, feeding, completion of food intake and tolerance diaries, reporting of AEs, and urine collection)
* Caregiver willing and able to sign IRB approved informed consent

Exclusion Criteria:

* Infant born with medical complications (e.g., neurological, cerebral palsy, etc.)
* Infant with failure to thrive, fever, any GI tract abnormalities (e.g., short gut, gastroesophageal reflux, etc.), any congenital illness or malformation that may affect infant feeding or normal growth
* Maternal, fetal, or infant medical history thought to have an impact on growth and/or development (substance abuse, positive HIV status, opioid exposure, or diabetes requiring insulin)
* Infant receiving prescription medication
* Infant with a known history of cow's milk protein allergy, excluding lactose intolerance
* Infant who has been treated with antibiotics or medications that may impact growth, GI tolerance and/or development
* Infant or family history (grandparent, parent, sibling) with known folate metabolism disorder
* Caregiver intent to feed non-study formula or solid food during the study

Ages: 0 Days to 11 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 394 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-07 (Actual)

PRIMARY OUTCOMES:
Weight Gain Velocity | Study Day 1 to Study Day 112
  Weight Gain Velocity (g/day)

SECONDARY OUTCOMES:
Length | Study Day 1 to Study Day 112
  Length and Length Gain Velocity (cm)
Head Circumference | Study Day 1 to Study Day 112
  Head Circumference and Head Circumference Gain Velocity (cm)
Formula Intake | Study Day 1 to Study Day 112
  Formula Intake Volume (oz/kg/day)
Formula Intake (2) | Study Day 1 to Study Day 112
  Formula Intake Volume (oz/day)
Anthropometry Z-scores | Study Day 1 to Study Day 112
  Weight for age Z-score, Length for age Z-score, Weight for length Z-score, Head circumference for age Z-score

OTHER OUTCOMES:
Adverse Event (AE) Assessment | Study Day 1 to Study Day 119
  AEs reported during the study
Caregiver report of stool consistency obtained during 3-consecutive day intervals | Study Day 1 to Study Day 112
  0=no bowel movement, 1=hard [dry hard pellets], 2=formed [definite shape, not dry], 3=loose [no definite shape, some water], 4=watery [no shape, mainly water])
Caregiver report of stool frequency obtained during 3-consecutive day intervals | Study Day 1 to Study Day 112
  Mean
Caregiver report of gassiness obtained during 3-consecutive day intervals | Study Day 1 to Study Day 112
  [a] Never [b] Rarely [c] Some of the time [d] Frequently [e] Always
Caregiver report of fussiness obtained during 3-consecutive day intervals | Study Day 1 to Study Day 112
  [a] Not at all [b] A little bit [c] Somewhat [d] Quite a bit [e] Very much
Caregiver report of spit up obtained during 3-consecutive day intervals | Study Day 1 to Study Day 112
  Mean
Caregiver report of crying obtained during 3-consecutive day intervals | Study Day 1 to Study Day 112
  Mean
Caregiver report of vomiting obtained during 3-consecutive day intervals | Study Day 1 to Study Day 112
  Mean
Urinalysis | Study Day 98 to Study Day 112
  Concentration of folate metabolites
Formula Satisfaction | Study Day 112
  Caregiver report using sliding scale of 1=Least to 5=Most

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lynch, MD, Principal Investigator — SPRIM Pro
Locations (1):
- SPRIM Pro, Indian Harbour Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided